CLINICAL TRIAL: NCT01838434
Title: A Phase I/Randomized Phase II Trial of Idelalisib and Lenalidomide in Patients With Relapsed/Refractory Mantle Cell Lymphoma
Brief Title: Lenalidomide With or Without Idelalisib in Treating Patients With Relapsed or Refractory Mantle Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Celgene Corporation (Industry); Gilead Sciences (Industry); Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A051201; NCI-2012-01734 (Registry Identifier: Clinical Trial Reporting Program); U10CA031946 (NIH)
Record Dates: First submitted 2013-04-19; First posted 2013-04-24 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Relapsed/Refractory Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Lenalidomide; idelalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lenalidomide (Phase II) (Active Comparator): Lenalidomide will be administered orally at 20 mg daily on days 1-21, repeated every 28 days for a maximum of 12 cycles (48 weeks). (Phase II)
  Interventions: Drug: lenalidomide
- lenalidomide and idelalisib (Phase II) (Experimental): Lenalidomide will be administered orally and daily on days 1-21, repeated every 28 days for a maximum of 12 cycles (48 weeks). Idelalisib will be orally administered for continuous 28-day cycles until progression, intolerance, or patient/physician discretion. Dosing will be determined by the Phase I portion of the study. (Phase II)
  Interventions: Drug: lenalidomide; Drug: idelalisib

INTERVENTIONS:
Drug: lenalidomide — given PO
Drug: idelalisib — given PO
  Arms: lenalidomide and idelalisib (Phase II)

SUMMARY:
This Phase I/II trial studies the safety and effectiveness of lenalidomide with or without idelalisib. Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Idelalisib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. It is not yet known whether lenalidomide is more effective with or without idelalisib in treating mantle cell lymphoma.

DETAILED DESCRIPTION:
A notice of temporary accrual suspension for Alliance A051201 was issued on 1/28/14. The study was suspended to new patient accrual until a protocol amendment was finalized, which provided revised treatment instructions. The study was reactivated on 4/22/14 including the removal of the rituximab treatment arm.

Outline: This is a phase I, dose-escalation study followed by a phase II study.

The phase I treatment plan includes the following:

1. Lenalidomide will be tested at sequential dose levels in a standard 3+3 design.

   1. Dose Level 0 = 15mg/day for days 1-21 every 28 days
   2. Dose Level 1 = 20mg/day for days 1-21 every 28 days and
   3. Dose Level 2 = 25mg/day for days 1-21 every 28 days.

   Patients can continue lenalidomide for up to 48 weeks (12 cycles) of treatment.
2. Idelalisib will be orally administered starting at 150 mg twice daily for continuous 28-day cycles until progression, intolerance, or patient/physician discretion. The dose is the same in dose levels 0, 1, and 2.

Patients are randomized to 1 of 2 treatment arms in the Phase II treatment plan. The primary and secondary objectives for this study are:

1. Phase I Primary Objective: To determine the safety and tolerability of the combination of lenalidomide with idelalisib in sequential dose cohorts.
2. Phase II Primary Objective: To determine the progression-free survival (PFS) of the combination of lenalidomide with or without idelalisib in a randomized phase II design.
3. Phase II Secondary Objectives:

   1. To determine the overall response rate (ORR), complete response rate (CR), and overall survival (OS) of the combination of lenalidomide with or without idelalisib in a randomized phase II design.
   2. To determine the prognostic and/or predictive significance of proliferation markers and cell cycle components in patients with relapsed/refractory mantle cell lymphoma (MCL) treated with idelalisib and lenalidomide.
   3. To determine whether phosphorylated protein kinase B (pAKT) expression levels are correlated with response to idelalisib plus lenalidomide.
   4. To determine whether Notch activation as assessed by notch homolog 1, translocation- association (NOTCH1) intracellular domain (ICD) immunohistochemistry (IHC) correlates with NOTCH1 mutational status and outcome in MCL patients treated with idelalisib and lenalidomide.
   5. To determine whether sex determining region Y-box 11 (SOX11) expression correlates with response in patients with relapsed/refractory MCL treated with idelalisib and lenalidomide.
   6. To correlate cereblon (CRBN) expression with response in patients with relapsed/refractory MCL treated with idelalisib and lenalidomide.
   7. To evaluate several plasma cytokines and correlate observed changes to objective response rates.

ELIGIBILITY:
1. Documentation of Disease:

   1. Histologically documented mantle cell lymphoma, with the following immunophenotypic characteristics: cluster of differentiation (CD)5+, (CD)23-, cyclin D1+; this may be from an initial diagnostic biopsy, or one obtained at time of relapse
   2. Institutional flow cytometry or immunohistochemistry must confirm CD5 antigen expression, lack of CD23 antigen expression, and expression of cyclin D1.
   3. Variant cases of mantle cell lymphoma will be eligible to participate after discussion and joint agreement between the PI, the Pathology Committee Chair, and the Lymphoma Committee Chair. Variant cases may include (but are not limited to) lack of Cyclin D1 expression (ie cases with Cyclin D2 or Cyclin D3 expression), CD23 negativity (if all other criteria are met), or alternative translocations leading to Cyclin D1 expression.
2. Prior Treatment - Patients must have prior treatment with at least one regimen, which may have been single agent or multi-agent, and consisted of traditional cytotoxic agents and/or biologic agents. Patient must not have received prior idelalisib or lenalidomide therapy. Patient must have progressive disease or refractory disease. Refractory disease will be defined as stable disease (SD) or progressive disease (PD) as best response to prior therapy.

   Progressive disease will be defined as complete response (CR) or partial response (PR) as initial response to prior therapy followed by disease progression within 6 months.

   Prior autologous, but not allogeneic, stem cell transplant is allowed. No corticosteroids within two weeks prior to study, except for maintenance therapy for a non-malignant disease. Maintenance therapy dose may not exceed 20 mg/day prednisone or equivalent.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status - Patients must have ECOG performance status of 0-2.
4. Measurable Disease must be present either on imaging studies. Non-measurable disease alone is not acceptable. Any tumor mass > 1 cm by computed tomography (CT), magnetic resonance imaging (MRI), or conventional radiograph is acceptable. Lesions that are considered non-measurable include the following:

   1. Bone lesions (lesions, if present, should be noted)
   2. Ascites
   3. Pleural/pericardial effusion
   4. Lymphangitis cutis/pulmonis
   5. Bone marrow (involvement by non-Hodgkin lymphoma should be noted)
5. Central Nervous System (CNS) Involvement - Patients must have no known CNS involvement by lymphoma.
6. Human Immunodeficiency Virus (HIV) Infection - Patients with HIV infection are eligible, provided they meet the following:

   1. CD4+ cell count > 350/mm3
   2. Treatment sensitive HIV and, if on anti-HIV therapy, HIV viral load < 50 copies/mm3
   3. No history of Acquired Immune Deficiency Syndrome (AIDS)-defining conditions or other HIV related illness
   4. No concurrent zidovudine or stavudine because of overlapping toxicities with protocol therapy
   5. Patients with known HIV positivity must have CD4 assessment and viral load at baseline and every 6 months while on study.
7. Pregnancy and Nursing Status - Patients must be non-pregnant and non-nursing. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10-14 days prior to registration. Further, they must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control: one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before starting lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP, even if they have had a successful vasectomy. A FCBP is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy, or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time preceding 24 consecutive months).
8. Deep Vein Thrombosis/Pulmonary Embolism (DVT/PE) - Patients with a recent history (within 3 months of study entry) of DVT/PE are not eligible. Patients with a distant history (greater than 3 months before study entry) of DVT/PE are eligible, but must receive either prophylactic aspirin or low molecular weight heparin, unless contraindicated.
9. Congestive Heart Failure - Patients must have no New York Heart Association (NYHA) Class III or Class IV congestive heart failure at study entry.
10. Myocardial Infarction - Patients must have no myocardial infarction within 6 months prior to study entry.
11. Hepatitis - Patients must not have known positivity for hepatitis B, as evidenced by + HBsAg or +anti-HBc, and must not have known history of hepatitis C.
12. Patients must be ≥ 18 years of age.
13. Cytochrome P450 3A4 (CYP3A4) Strong Inducers and Inhibitors - Patients must not be on strong CYP3A4 inhibitors and/or inducers.

    1. The following strong inhibitors are prohibited: indinavir, nelfinavir, ritonavir, clarithromycin, itraconazole, ketoconazole,nefazodone
    2. The following strong inducers are prohibited: carbamazepine, phenobarbital, phenytoin, pioglitazone, rifabutin, rifampin, St. John's Wort, troglitazone
14. Required Initial Laboratory Values:

    1. ANC ≥ 1,000/µL, ≥ 500/µL if marrow involvement
    2. Platelets ≥ 75,000/µL
    3. Creatinine ≤ 1.5 x ULN, and estimated creatinine clearance ≥ 60 mL/min (patients on dialysis not eligible), unless attributable to non-Hodgkin lymphoma
    4. Total bilirubin ≤ 2 x ULN, unless attributable to non-Hodgkin lymphoma or Gilbert's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09-30 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of idelalisib and lenalidomide, determined according to incidence of dose-limiting toxicity (DLT) graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (Phase I) | 28 days
Progression Free Survival (PFS) of the combination of lenalidomide, with or without idelalisib (Phase II) | Time between registration and disease progression or death, assessed up to 2 years

SECONDARY OUTCOMES:
Overall survival (OS) (Phase II) | Up to 2 years
Overall response rate (partial or complete response) (Phase II) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sonali Smith, MD, Study Chair — University of Chicago
Locations (4):
- United States (4):
  - University of Chicago, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Ohio State University Medical Center, Columbus, Ohio

REFERENCES:
- [Derived] Smith SM, Pitcher BN, Jung SH, Bartlett NL, Wagner-Johnston N, Park SI, Richards KL, Cashen AF, Jaslowski A, Smith SE, Cheson BD, Hsi E, Leonard JP. Safety and tolerability of idelalisib, lenalidomide, and rituximab in relapsed and refractory lymphoma: the Alliance for Clinical Trials in Oncology A051201 and A051202 phase 1 trials. Lancet Haematol. 2017 Apr;4(4):e176-e182. doi: 10.1016/S2352-3026(17)30028-5. Epub 2017 Mar 15. PMID 28314699